CLINICAL TRIAL: NCT03929094
Title: A Phase II, Single-arm Study to Evaluate the Efficacy and Safety of the Combination of Nab-paclitaxel and Gemcitabine in Treating Patients With Metastatic Pancreatic Cancer
Brief Title: Nab-paclitaxel and Gemcitabine in Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-22
Record Dates: First submitted 2019-03-15; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel + gemcitabine (Experimental): nab-paclitaxel at 100 mg/m^2 on days 1, 8, and 15; gemcitabine at 1000 mg/m^2 on days 1, 8, and 15
  Interventions: Drug: Paclitaxel for Injection（Albumin Bound）; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel for Injection（Albumin Bound） — Patients firstly receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic.
  Other Names: Paclitaxel
Drug: Gemcitabine — Patients secondly receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic.

SUMMARY:
This is a single arm, open-label Phase II clinical trial to Evaluate the Efficacy and Safety of the Combination of Nab-paclitaxel and Gemcitabine in Treating Patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
While GT (Gemcitabine + Nab-paclitaxel) is one of the preferred regimens for metastatic pancreatic cancer, we have yet to determine the optimum number of cycles for GT treatment regimen. In this single arm, open-label clinical trial, metastatic pancreatic cancer patients will be received nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) and gemcitabine 1000 mg/m^2 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel therapeutic.

The safety and efficacy of each group will be assessed through ORR, PFS, OS and adverse effects as graded by CTC-AE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed content obtained prior to treatment. The patients were fully explained and understood the purpose, contents, predicted efficacy, pharmacological effects, and risks of this study.
2. target population

   * the patients were confirmed as metastatic pancreatic cancer by histopathology or cytopathology.
   * At least one measurable objective lesion (both primary and metastatic) was identified based on the RECIST1.1 criteria;
   * Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
   * The expected survival after surgery ≥ 3 months
   * The subjects have good compliance, can be treated and followed up, and voluntarily comply with the relevant provisions of this study
   * No contraindications for gemcitabine and nab-paclitaxel.
3. Age and reproductive status

   * Age ≥ 18 years and ≤ 75 years
   * Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age 24 hours before the start of chemotherapy;
   * Women must not lactate.

Exclusion Criteria:

1. The target disease has cerebral metastasis;
2. medical history and complications

   * patients had uncontrolled serious medical condition that the investigator considered may affect the subject's to receive treatment under the study program, For example, patients with severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
   * Dementia, changing of mental state or any mental illness which could hinder understanding or informed consent or fill out questionnaires;
   * History of allergy or hypersensitivity to any therapeutic ingredient;
   * Combined with other malignant tumors excepted pancreatic cancer within the first 5 years of randomization, excepted well-treated basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical resection, and ductal carcinoma in situ of the breast after radical resection.
   * Previously received systemic therapy for advanced/metastatic pancreatic cancer;
   * Subjects who had previously been pathologically diagnosed with squamous cell carcinoma (no organ limitation) and received neoadjuvant/adjuvant therapy with taxa regimen.
   * Patients who had Grade 2 or above Peripheral neuropathy.
3. Abnormal results of physical examination and laboratory examination

   * Absolute neutrophil count (ANC) 90g/L 1.5 × 109/L; Platelets (PLT) 90g/L 100 × 109/L; Hemoglobin (Hgb) < 90g/L
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) >2.5 × institutional upper limit of normal (ULN), >5 × institutional upper limit of normal (ULN) (hepatic metastases); Total bilirubin (TBIL)>1.5 × ULN;
   * Creatinine (CRE)> 1.5 × ULN
   * Prothrombin time (PT) and international normalized ratio (INR) > 1.5 × ULN. Unless the subject had received anticoagulant treatment
4. Subjects had hepatitis b surface antigen (HBsAg)-positive and hbv-dna titer in peripheral blood greater than or equal to 1000 copy number /L;If HBsAg is positive and the peripheral blood hbv-dna <1000 copy number /L, the subjects will be eligible for inclusion if the investigator considers that chronic hepatitis b is stable and does not increase the risk of subjects.
5. Human immunodeficiency virus (HIV)- or hepatitis C virus (HCV) positive patients;
6. Patients combined with other anti-tumor drugs.
7. Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period.
8. The researchers considered that there were other conditions that were not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | through study completion, an average of 1 year
  To evaluate the Overall Response Rate of patients with metastatic pancreatic cancer after treated with nab-paclitaxel plus gemcitabine.
Progression Free Survival | through study completion, an average of 1 year
  To evaluate the Progression Free Survival of patients with metastatic pancreatic cancer after treated with nab-paclitaxel plus gemcitabine.

SECONDARY OUTCOMES:
overall survival | through study completion, an average of 1 year
  To evaluate the overall survival of patients with metastatic pancreatic cancer after treated with nab-paclitaxel plus gemcitabine.
adverse events | through study completion, an average of 1 year
  adverse events of patients with metastatic pancreatic cancer after treated with nab-paclitaxel plus gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, Study Director — Fudan University
Locations (1):
- FUDAN University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No